CLINICAL TRIAL: NCT02238314
Title: Tipranavir Disodium: An Open-Label ExploratorySstudy of Tipranavir and Ritonavir in Combination With One Nucleoside Reverse Transcriptase Inhibitor and One Non-Nucleoside Reverse Transcriptase Inhibitor in Multiple Protease Inhibitor-Experienced HIV Patients
Brief Title: Exploratory Study of Tipranavir and Ritonavir in Multiple Protease Inhibitor-experienced HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.2
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

ARMS (2):
- Tipranavir low dose (Experimental)
  Interventions: Drug: Tipranavir low dose; Drug: Ritonavir; Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTI); Drug: Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI)
- Tipranavir high dose (Experimental)
  Interventions: Drug: Tipranavir high dose; Drug: Ritonavir; Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTI); Drug: Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI)

INTERVENTIONS:
Drug: Tipranavir low dose
  Arms: Tipranavir low dose
Drug: Tipranavir high dose
  Arms: Tipranavir high dose
Drug: Ritonavir
Drug: Nucleoside Reverse Transcriptase Inhibitor (NRTI)
Drug: Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI)

SUMMARY:
The primary objective was to evaluate the antiviral activity and safety of two regimens of tipranavir (500 mg BID or 1000 mg BID) plus ritonavir (100 mg BID) administered in combination with 1 new nucleoside reverse transcriptase inhibitor (NRTI) + efavirenz in multiple protease-inhibitor-experienced HIV-1 positive patients.

ELIGIBILITY:
Inclusion Criteria:

* Multiple (two or more) PI-experience. Eligible patients must have had exposure to at least two antiretroviral regimens containing a single protease inhibitor or a regimen containing dual protease inhibitors
* In the investigator's opinion, the patient had adhered to PI-containing regimens
* Exposure of ≥ 3 months to the current PI therapy
* Exposure of ≥ 4 months to the prior PI therapy with single PI-containing regimens
* Stable PI-containing regimen for at least 2 months prior to study entry
* HIV-1-RNA ≥ 5,000 copies/mL
* Cluster of differentiation (CD)4+ cell count ≥ 50 cells/mm**3
* At least one new NRTI option available
* Age ≥ 13 years
* Acceptable screening laboratory values that indicated adequate baseline organ function at the time of screening. Laboratory values were considered acceptable if the severity was ≤ Grade 1 (AIDS Clinical Trial Group (ACTG) Grading Scale). Stable Grade 2 abnormalities were permitted if the values had been demonstrated and documented for at least ≥ 2 months.
* Acceptable medical history, physical examination, electrocardiogram, and chest X-ray prior to entry into the treatment phase of the study
* Agreement to use a barrier contraceptive method of birth control for at least 30 days prior to study drug administration, during the study, and 30 days after the end of the study
* Ability to swallow numerous tablets and capsules without difficulty
* Ability to understand and provide informed consent. Minors were required to have approval of a parent or legal guardian

Exclusion Criteria:

* Prior exposure, defined as > 7 treatment days, to nonnucleoside reverse transcriptase inhibitor (NNRTIs) including, but not limited to: nevirapine, efavirenz, delavirdine, atevirdine, MKC-442, loviride, and HBY-097
* Clinically significant active or acute (onset within the month previous to study entry) medical problems, including the following: opportunistic infections, such as active cryptococcosis, Pneumocystis carinii pneumonia, herpes zoster, histoplasmosis, or cytomegalovirus or nonopportunistic diseases, including, but not limited to, progressive multifocal leukoencephalopathy, lymphoma, or malignancy requiring systemic therapy
* Prior exposure (> 7 days) to tipranavir
* History of clinically significant nervous system or muscle diseases, seizure disorder, or psychiatric disorder that might impair adherence to the protocol
* Taking of any known P450 3A enzyme-inducing drugs within 30 days of study entry and including the following: rifabutin, rifampin, carbamazepine, dexamethasone, phenobarbital, phenytoin, sulfadimidine, sulfinpyrazone, or troleandomycin
* Hypersensitivity to tipranavir and/or ritonavir
* Use of interferons, interleukins, HIV vaccines, or any active immunizations within 30 days prior to study entry
* Taking of any investigational medication with the exception of adefovir dipivoxil (Preveon™) and amprenavir (Agenerase™) within 30 days of study entry
* Pregnancy or lactation (serum β-human chorionic gonadotrophin test had to have been negative within 14 days of study entry)
* Evidence of active substance abuse, which in the investigator's opinion, could affect compliance to the protocol
* In the investigator's judgment, inability to comply with the protocol requirements for reasons other than those specified

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1999-01; Primary Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HIV-1 RNA concentrations | weeks 16, 24, 48 and 80
Occurrence of HIV-1 RNA levels below the limit of quantitation (BLQ) (400 copies/mL) | up to 112 weeks
  measured by the Roche Amplicor HIV-1 Monitor™ polymerase chain reaction (PCR) Method
Occurrence of HIV-1 RNA levels BLQ (50 copies/mL) | up to 112 weeks
  measured by the Roche Amplicor UltraSensitive™ PCR Method
Number of patients with treatment-emergent and drug-related adverse events (AEs) | up to 115 weeks
Number of patients with serious adverse events (SAEs) | up to 115 weeks
Number of patients with grade 3 and 4 laboratory abnormalities | up to 115 weeks

SECONDARY OUTCOMES:
Change from baseline in cluster of differentiation (CD) 4+ cell count responses | weeks 24, 48 and 80
Change from baseline in CD8+ cell count responses | weeks 24, 48 and 80
Time to new or recurring AIDS-defining illness | up to 115 weeks
Time to new or recurring HIV-related illness | up to 115 weeks
Time to death | up to 115 weeks
Occurrence of AIDS-defining illness, | up to 115 weeks
Occurrence of HIV-related illness, | up to 115 weeks
Occurrence of death | up to 115 weeks
Time to virologic failure | up to 115 weeks
  defined as plasma HIV-1 RNA values >400 copies/mL or a 0.5 log reduction from baseline at two consecutive time points
Change from baseline in cholesterol | up to 115 weeks
Change from baseline in HDL | up to 115 weeks
Change from baseline in triglycerides | up to 115 weeks
Change from baseline in blood glucose | up to 115 weeks
Steady-state plasma concentrations | up to week 24
Fold-change in concentration required to produce 50% of inhibition (IC 50) | Baseline, weeks 24, 48 and 80
  sequence-based HIV-1 analysis (genotyping) and drugs susceptibility assays (phenotyping)